CLINICAL TRIAL: NCT05514158
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Disitamab Vedotin Combined With RC98 in the Treatment of Subjects With HER2-expressing Locally Advanced or Metastatic Gastric Cancer (Including AEG).
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Disitamab Vedotin Combined With RC98 in the Treatment of Subjects With HER2-expressing Locally Advanced or Metastatic Gastric Cancer (Including AEG)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C015
Record Dates: First submitted 2022-08-04; First posted 2022-08-24 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 combind with RC98 (Experimental)
  Interventions: Drug: RC48-ADC; Drug: RC98

INTERVENTIONS:
Drug: RC48-ADC — RC48 for injection is a novel antibody-drug conjugate, with a her-2-targeting antibody and a microtube inhibitor
  Other Names: RC48-ADC injection
Drug: RC98 — RC98 is a recombinant humanized IgG1 monoclonal antibody targeting programmed cell death-Ligand 1 (PD-L1)
  Other Names: RC98 injection

SUMMARY:
This is a single-center, open-label, dose-escalation phase I clinical study.This study aimed to evaluate the safety, tolerability, pharmacokinetics and preliminary clinical efficacy of RC48-ADC combined with RC98 in subjects with advanced gastric cancer.Which will provide a reference basis for dose confirmation in subsequent clinical studies.

DETAILED DESCRIPTION:
The dose escalation phase will enroll subjects with HER2-expressing locally advanced or metastatic gastric cancer, including gastroesophageal junction adenocarcinoma. HER2 expression is defined as follows (meets one of the following):

• HER2 IHC3+, 2+, 1+; (Subjects with HER2 immunohistochemistry (IHC) results of IHC1+, IHC 2+, and IHC 3+, previous test results (confirmed by the investigator) or research center test results are acceptable;

The dose-escalation phase preset doses for this combination therapy are as follows:

RC48-ADC: 2.5mg/kg Q2W; RC98 increasing dose: 5.0mg/kg Q2W, 10.0mg/kg Q2W, 15.0mg/kg Q2W. The dose escalation phase of the combination therapy adopts the Bayesian optimal interval (BOIN) design method: the fixed dose of RC48-ADC is 2.5 mg/kg, and the dose of RC98 is escalated, and the initial incremental dose of RC98 is 5.0 mg/kg. MTD has a target toxicity rate of 0.3 and a maximum sample size of 24. The subjects will be enrolled in units of 3, with a maximum of 12 subjects in each dose group; the 28 days after the first dose will be used as the observation window of DLT to make decisions such as dose increase and decrease. If the DLT criteria were not met within 28 days after the first dose, dose escalation was not continued to observe DLT and MTD. After the dose escalation period is over, the investigator decides the recommended phase 2 dose (RP2D) based on the available safety, tolerability, PK, and efficacy information.

After completing the dose-limiting toxicity (DLT) evaluation, the subject can continue to receive the original dose of study drug treatment (but not more than the currently ongoing escalating dose or the maximum tolerated dose under the condition that the investigator judges that there may be benefits) ), subjects received treatment until intolerable toxicity, disease progression, or termination of the study by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the research and sign the informed consent;
2. Age 18-70 (including 18 and 70);
3. Expected survival period ≥ 12 weeks;
4. ECOG performance status of 0 or 1 within 3 days before the first dose of study treatment;
5. Patients with metastatic or unresectable locally advanced or metastatic gastric cancer (including gastroesophageal junction adenocarcinoma) confirmed by histology or cytology with disease progression after standard treatment or intolerant to standard treatment;
6. Female subjects should be surgically sterilized, postmenopausal patients, or agree to use at least one medically approved contraceptive measure (such as an intrauterine device, contraceptives) during the study treatment period and within 6 months after the end of the study treatment period. pills or condoms), must have a negative blood pregnancy test within 7 days prior to study enrollment, and must be non-nursing. Male subjects should agree to use at least one medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period;
7. Able to understand trial requirements, willing and able to comply with trial and follow-up procedures.

Adequate organ and bone marrow hematopoiesis 8. Bone marrow function:

* Hemoglobin≥90g/L;
* Absolute neutrophil count ≥1.5×109/L;
* Platelets≥100 × 109/L; 9. Liver function (subject to the normal value of the clinical trial center):
* In the absence of liver metastases, the total serum bilirubin is ≤1.5 times the ULN; in the presence of liver metastases, the total serum bilirubin is ≤3 times the ULN;
* In the absence of liver metastases, both ALT and AST are ≤3 times ULN, and in the presence of liver metastases, both ALT and AST are ≤5 times ULN; 10. Renal function (subject to the normal value of the clinical trial center):
* Serum creatinine ≤ 1.5 times ULN, or creatinine clearance (CrCl) ≥ 60 mL/min calculated by the Cockcroft-Gault formula, or 24-hour urine CrCl ≥ 60 mL/min; 11. Coagulation function: International normalized ratio (INR), activated partial thromboplastin time (APTT) and prothrombin time (PT) are all ≤1.5 times ULN; 12. Endocrine function: Thyroid-stimulating hormone (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) are within the normal range of ±10%; 13. Heart function:
* New York Heart Association (NYHA) class <3;
* Left ventricular ejection fraction ≥50%; 14. At least one measurable lesion according to RECIST 1.1 criteria; 15. The HER2 IHC test results are IHC 1+, IHC 2+ or IHC 3+, the subject's previous test results (confirmed by the investigator) or the test results of the research center are acceptable, and can provide a diagnosis of locally advanced or metastatic gastric cancer of tumor tissue specimens, as well as a sufficient number of paraffin blocks, tissue sections (5-10 unstained) for biomarker detection.

Exclusion Criteria:

1. The study drug has been used within 4 weeks before the start of the study drug;
2. Major surgery has been performed within 4 weeks before the start of the study drug and the patient has not fully recovered;
3. Have been vaccinated with live vaccines within 4 weeks before the start of the study drug or plan to receive any vaccines during the study period (except for the new coronavirus vaccine);
4. Arterial/venous thrombotic events, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism, occurred within 6 months before the study drug;
5. Major cardiovascular disease (NYHA grade 3 or 4 heart failure, second-degree or higher heart block, myocardial infarction within the past 12 months, unstable arrhythmia or unstable angina pectoris, cerebral infarction within 6 months infarction, etc.);
6. Active autoimmune disease requiring systemic treatment (such as the use of immunomodulatory drugs, corticosteroids or immunosuppressants) within 2 years before the start of study administration, allowing related replacement therapy (such as thyroxine, insulin, or renal or Physiological corticosteroid replacement therapy for pituitary insufficiency);
7. Subjects who need to receive glucocorticoid (prednisone>10 mg/day or other similar drugs at an equivalent dose) or other immunosuppressive therapy due to certain conditions within 14 days before the start of the study drug;
8. Suffering from uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, liver cirrhosis, etc.;
9. Suffering from active infection requiring systemic treatment;
10. History of active tuberculosis;
11. Positive human immunodeficiency virus (HIV) test result;
12. Hepatitis B surface antigen (HBsAg) positive and HBV DNA copy number greater than the upper limit of the normal value of the laboratory department of the research center; or hepatitis C virus (HCV) antibody positive and the HCV RNA copy number greater than the upper limit of the normal value of the laboratory department of the research center;
13. Conditions that the investigator believes will affect the safety or compliance of the drug treatment in this study, including but not limited to moderate to large amounts of pleural/ascites/pericardial effusion, difficult-to-correct pleural/ascites/pericardial effusion, mental illness, etc.;
14. Known to have hypersensitivity reactions or delayed allergic reactions to certain components of RC98 for injection or similar drugs;
15. Those who are known to be allergic to recombinant humanized anti-HER2 monoclonal antibody-MMAE conjugate drugs and their components;
16. Previously received PD-(L)1 inhibitor or other antibody-conjugated drug therapy;
17. Suffering from any other disease, metabolic abnormality, abnormal physical examination or abnormal laboratory test, according to the judgment of the investigator, there is reason to suspect that the subject has a certain disease or condition that is not suitable for the use of the study drug, or will affect the research results interpretations, or situations that place the subject at high risk;
18. Women who are pregnant or breastfeeding or women/men who are planning to give birth;
19. It is estimated that the subjects' compliance to participate in this clinical study is insufficient or the investigators believe that there are other factors that are not suitable for participating in this study; tumor related
20. Suffering from central nervous system metastases and/or cancerous meningitis. Subjects who have previously received treatment for brain metastases may be considered for participation in this study, provided that their disease has been stable for at least 3 months, no disease progression has been confirmed by imaging within 4 weeks prior to the first dose of the study, and all neurological symptoms have recovered At baseline, there was no evidence of new or enlarging brain metastases, and radiation, surgery, or steroid therapy was discontinued at least 28 days prior to the first dose of study treatment. This exception does not include cancerous meningitis, which should be excluded regardless of its clinically stable status;
21. Suffering from other malignant tumors within 5 years before signing the informed consent form (non-melanoma skin cancer, cervical carcinoma in situ or other tumors that have been effectively treated, except for malignant tumors that are considered cured);
22. Received chemotherapy and radiotherapy within 4 weeks before the start of the study drug;
23. Subjects who have received immune-enhancing therapy (such as alpha-interferon, interleukin-2) within 2 weeks before the start of the study drug.
24. Received hormone therapy for the tumor within 2 weeks before the start of the study drug;
25. Received palliative radiotherapy for bone metastases within 2 weeks before the start of the study drug;
26. Received anti-tumor traditional Chinese medicine treatment within 2 weeks before the start of the study drug;
27. The toxicity caused by previous anti-tumor therapy has not recovered to CTCAE (version 5.0) grade 0-1 (except for 2nd degree alopecia);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after first treatment
  In the DLT evaluation window (observation period 1-28 days after the first administration), according to the NCI-CTCAE v5.0 grading standard, the investigator or the sponsor believes that toxic reaction which are reasonably related to RC48 and/or RC98 treatment
The incidence and severity of adverse events (AE) | From the day of ICF sign to 28 days after the day of the last treatment
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Cmax of RC48 | 24 months
  Peak Plasma Concentration of RC48
AUC of RC48 | 24 months
  Area under the plasma concentration versus time curve of RC48
Cmax of RC98 | 24 months
  Peak Plasma Concentration of RC98
AUC of RC98 | 24 months
  Area under the plasma concentration versus time curve of RC98
AUC of MMAE | 24 months
  Area under the plasma concentration versus time curve of MMAE
Cmax of MMAE | 24 months
  Peak Plasma Concentration of MMAE
Immunogenicity of RC48 | 24 months
  Anti-drug antibody (ADA) of RC48 positive samples, etc.
Immunogenicity of RC98 | 24 months
  Anti-drug antibody (ADA) of RC98 positive samples, etc.
Objective response rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Duration of Remission (DOR) | 24 months
  Duration of response is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Disease Control Rate(DCR) | 24 months
  Proportion of patients whose tumors shrank or stabilized for a certain period of time
Progression-free survival | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions

CONTACTS AND LOCATIONS:
Overall Officials: yi Ba, ph.D, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Remegen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No